CLINICAL TRIAL: NCT01637545
Title: Phase 4 Study of Nasea(R)/Ramosetron Inj.as Anti-emetics in the Patients Undergoing Facial Bone Fracture Operations
Brief Title: Evaluation of Safety and Efficacy of Nasea(R)/Ramosetron Inj. in Patients Undergoing Facial Bone Fracture Operations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator is away on business
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Yeong Heo, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1107-131-007; L-2011-329-1 (Other Grant/Funding Number: Astellas Pharm. Co.)
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Facial Bones Fracture
Keywords: facial bones; Post operative nasea vomiting; fractures; reduction
MeSH Terms: conditions — Fractures, Bone | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Preop. ramosetron 0.3mg i.v. (Active Comparator): G1 - Ramosetron 0.3mg i.v. just before the beginning of the surgery
  Interventions: Drug: Ramosetron
- Postop. ramosetron 0.3mg i.v. (Active Comparator): G2 - Ramosetron 0.3mg i.v. just after the end of the surgery and moving into the Recovery room
  Interventions: Drug: Ramosetron
- No Ramosetron (Active Comparator): G3 - No medication but regular antiemetics injection if the patient wants
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — G1 - Ramosetron 0.3mg i.v. just before the beginning of the surgery G2 - Ramosetron 0.3mg i.v. just after the end of the surgery and moving into the Recovery room
  G3 - No medication but regular antiemetics injection if the patient want
  Other Names: Nasea®

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most common and distressing complications after anaesthesia and surgery, and may lead to serious postoperative complications This prospective, randomized study designed to evaluate the best injection time to get the prophylactic anti-emetic efficacy of ramosetron, a newly developed 5-HT(3) antagonist in patients undergoing facial bone surgery.

DETAILED DESCRIPTION:
1. Participants

   * 100 patients with undergoing facial bone surgery are going to be randomly allocated to one of the 3 groups
2. Randomization

   * G1(n=33) - Ramosetron 0.3mg i.v. just before the beginning of the surgery
   * G2(n=33) - Ramosetron 0.3mg i.v. just after the end of the surgery and moving into the Recovery room
   * G3(n=33) - No medication but regular antiemetics i.v. if the patient wants
3. The primary endpoint

   * the incidence of nausea and vomiting for 24 h after surgery at 0-6h, 6-12 h and 12-24 h
4. The secondary endpoints

   * the severity of nausea, need for rescue medication
   * patient satisfaction with efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patient who sign informed consent form for the study
* patient who are considered as surgical candidates with facial bones fracture

Exclusion Criteria:

* Patient who have had nausea/vomiting episodes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
incidence and severity of nausea and vomiting | for 24 h after surgery at 0-6h, 6-12 h and 12-24 h

SECONDARY OUTCOMES:
patient satisfaction with the effect | at 24 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea